CLINICAL TRIAL: NCT03777514
Title: A Randomized, Placebo-controlled Comparator Trial of IV vs Oral Iron Treatment of Iron Deficiency Anemia in the Post-operative Bariatric Surgical Patient
Brief Title: Intravenous (IV) Versus Oral Iron Treatment of Iron Deficiency Anemia in the Post-operative Bariatric Surgical Patient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study wasn't started.
Sponsor: Johns Hopkins University (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00198735
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: IDA in the Post-bariatric Surgical Patient
MeSH Terms: interventions — Ferrosoferric Oxide; ferrous sulfate; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The study is a randomized, comparative double blind, double dummy study to evaluate efficacy and time course of treatment response of bariatric surgical patients found to have IDA, three months or greater following bariatric surgery (Roux-en Y gastric bypass and vertical sleeve gastrectomy) over 6 weeks with a 46-week follow-up extension. Two medications and placebos will be used with equal random assignment to both groups
  * Ferumoxytol intravenous (IV) 1020 mg as - 2 vials of 510 mg (510 mg IV over 15 minutes) each given 2-7 days apart.
  * Ferrous sulfate 325 mg (oral) tabs morning and evening.
  * Placebo: oral vitamin C 500 mg tabs, saline infusion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IV bags will be opaque and patients will be asked to wear a eye mask during the infusion of iron vs. saline.
  The oral tables will be identical in color and shape (iron in the form of ferrous sulphate and vitamin C)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV iron (Active Comparator): Ferumoxytol intravenous (IV) 1020 mg as - 2 vials of 510 mg (510 mg IV over 15 minutes) each given 2-7 days apart.
  Participants in this group will also receive oral vitamin C as a placebo.
  Interventions: Drug: Ferumoxytol; Other: Oral vitamin C
- oral iron (Active Comparator): Ferrous sulfate 325 mg (oral) tabs morning and evening. Participants in this group will also receive intravenous normal saline as a placebo.
  Interventions: Drug: Ferrous sulfate; Other: Intravenous normal saline

INTERVENTIONS:
Drug: Ferumoxytol — treatment of iron deficiency anemia with IV iron.
  Arms: IV iron
Drug: Ferrous sulfate — treatment of iron deficiency anemia with oral iron
  Arms: oral iron
Other: Oral vitamin C — Oral vitamin C to be used as a placebo for participants receiving IV iron
  Arms: IV iron
Other: Intravenous normal saline — Intravenous normal saline will be used as placebo for participants receiving oral iron
  Arms: oral iron

SUMMARY:
The aim of the study is to compare two accepted treatments for iron deficiency anemia (oral ferrous sulfate and intravenous ferumoxytol) for efficacy and speed of response in the treatment of iron deficiency anemia (IDA) in the post-operative bariatric surgical patient. In this study, 104 bariatric surgical post-operative patients will be randomly assigned 52 each to oral or 52 to a single dose IV iron treatment using double-blind procedures.

DETAILED DESCRIPTION:
Rationale for study: The preponderance of published evidence reports superior efficacy and decreased toxicity of intravenous iron compared to oral iron in correcting anemia and iron parameters in published trials of bariatric surgery patients. Intravenous, and not oral, iron ensures adequate delivery and avoids gastrointestinal toxicities, which may be especially burdensome in these patients who require optimal levels of energy to maintain prudent exercise programs recommended by patients' bariatric practitioners. Uncontradicted published evidence reports safety and efficacy of complete replacement doses of intravenous iron administered in one or two doses of either low molecular weight iron dextran, ferumoxytol, ferric carboxymaltose or iron isomaltoside. A common feature of all studies extant is the lack of reported serious adverse events. Even in patients with minimally invasive procedures such as gastric banding or stapling in whom oral iron may be tolerated, given the often present multiple gastrointestinal perturbations, intravenous iron may simplify care.

Drugs used: The investigators propose to use and FDA approved IV iron preparation - ferumoxytol, administered as two doses (over a interval of 2 to 7 days), each 510 mg over fifteen minutes based on published prospective safety and efficacy data and compare the effectiveness of the treatment to the American Metabolic and Bariatric Associations recommended treatment for iron deficiency anemia in the post-operative bariatric patients of oral iron ferrous sulphate 325 mg twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Patients who have undergone a Roux-en Y Gastric Bypass or Vertical Sleeve Gastrectomy and are at least 3 months or more out from surgery.
* Iron deficiency anemia defined as iron deficient with either ferritin < 20 mcg/l, transferrin saturation (TSAT) < 19%, or anemia with Hgb < 13 g/dL for both males and females.
* Willingness to use contraceptive to avoid pregnancy: Women have to be surgically sterile, post menopausal or use one of the following contraceptives during the whole study period and after the study has ended for at least five times the plasma biological half-life of the investigational medicinal product: intrauterine devices or hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release).
* Willingness to participate and signing the informed consent form.

Exclusion Criteria:

* Iron overload or disturbances in utilization of iron (e.g. hemochromatosis and hemosiderosis)
* Decompensated liver cirrhosis or active hepatitis (ALT > 3 times upper limit of normal)
* Serum ferritin > 500 ng/mL or transferrin saturation > 40%
* Active acute or chronic infections (assessed by clinical judgment that may be indicated by White Blood Cells (WBC) and C-Reactive Protein (CRP) when these are available)
* Rheumatoid arthritis with symptoms or signs of active inflammation
* Pregnant and nursing women
* History of multiple allergies
* Known hypersensitivity to ferumoxytol or oral iron or any excipients in the drug products
* Previous IV iron treatment for IDA
* Other iron treatment or blood transfusion within 4 weeks prior to the screening or treatment visit
* Planned elective surgery during the study
* Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study, e.g. a malignancy, uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Resolution of anemia in oral vs. IV iron as assessed by Clinical Global Impression (CGI) - 2 score | 6 weeks
  The CGI-2 is a one-item questionnaire which asks how participants feel now compared to before receiving treatment. It has a scoring of 1 to 7 with 1 meaning much better and 7 meaning very much worse
Resolution of anemia in oral vs. IV iron as assessed by ferritin level | 6 weeks
  Participants will be assessed after six weeks to see if there is a resolution of anemia following the treatment with oral or IV iron. This will be determined by the ferritin level. Ferritin > 20% will be the cutoff for resolution of anemia.
Resolution of anemia in oral vs. IV iron as assessed by TSAT | 6 weeks
  Participants will be assessed after six weeks to see if there is a resolution of anemia following the treatment with oral or IV iron. This will be determined by TSAT level. TSAT > 19% will be the cutoff for resolution of anemia.
Time (weeks) to treatment response as assessed by CGI-2 score | 6 weeks
  The CGI-2 is a one-item questionnaire which asks how participants feel now compared to before receiving treatment. It has a scoring of 1 to 7 with 1 meaning much better and 7 meaning very much worse. This will be used in assessing the time in weeks when participant noticed a change after receiving treatment.
Time (weeks) to treatment response as assessed by ferritin level | 6 weeks
  Participants will be assessed after six weeks to identify what time (in weeks) ferritin level was > 20% following the treatment with oral or IV iron
Time (weeks) to treatment response as assessed by TSAT | 6 weeks
  Participants will be assessed after six weeks to identify what time (in weeks) TSAT level was > 19% following the treatment with oral or IV iron

SECONDARY OUTCOMES:
Need for continued treatment as assessed by ferritin level | 1 year
  Participants will be assessed after a year to see if participants require continued treatment following the treatment with oral or IV iron. This will be determined by the ferritin level. Ferritin > 20% will be the cutoff for no further need for treatment.
Need for continued treatment as assessed by TSAT | 1 year
  Participants will be assessed after a year to see if participants require continued treatment following the treatment with oral or IV iron. This will be determined by TSAT level. TSAT > 19% will be the cutoff for no further need for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley E Steele, MD, Ph.D, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No